CLINICAL TRIAL: NCT01193816
Title: Assessment of Loxapine in the Management of Restlessness During Mechanical Ventilation Weaning
Brief Title: Loxapine in the Management of Restlessness During Mechanical Ventilation Weaning
Acronym: Sevralox
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P 070106
Record Dates: First submitted 2010-08-26; First posted 2010-09-02 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Restlessness
Keywords: restlessness during mechanical ventilation weaning
MeSH Terms: conditions — Psychomotor Agitation | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- loxapine (Experimental): loxapine
  Interventions: Drug: loxapine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: loxapine — Each patient may receive a maximum dosage of 900mg of Loxapine per day (drinkable solution through gastric probe) or the same volume of placebo. 2 initial administrations of 150 mg followed by potential readministration of 100 mg of loxapine. Maximum duration of treatment will be 14 days.The dosage by day is defined by patients' clinical condition, assessed with RASS score.
  Arms: loxapine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to assess the efficacy of a drug (loxapine, a neuroleptic) in calming patients down in a situation of restlessness during mechanical ventilation weaning. This drug is used for several years to quieten restless patients. Its purpose is to restore spontaneous breathing sooner and therefore to reduce the risks of intubation and mechanical ventilation.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of a drug (loxapine, a neuroleptic) in calming patients down in a situation of restlessness during mechanical ventilation weaning. This drug is used for several years to quieten restless patients. Its purpose is to restore spontaneous breathing sooner and therefore to reduce the risks of intubation and mechanical ventilation. 300 patients will participate in the study and will be randomized, after informed consent, to receive either loxapine or a placebo.Patients whose proxies refuse participation will be sedated according to standard care procedures.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* sedated
* under mechanical ventilation through intubation probe for more than 48 hours
* no contra-indication to naso-gastric probe- with criteria for potential weaning
* with social security
* important restlessness at sedation withdrawal, defined as RASS score (Richmond Agitation Sedation Scale)= 2. This restlessness has no potential danger for the patient but requires a level of sedation. This re-sedation implies administration of morphinomimetics and benzodiazepines at dosages that does not allow to pursue mechanical ventilation weaning attempts.

Exclusion Criteria:

* extreme restlessness at sedation withdrawal ((RASS>2)
* allergy to loxapine or one of its component
* dopaminergic agonists
* extubation planned in the following 24 hours
* antecedent of comitiality
* known pregnancy at admission
* proxies opposed to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Weaning period | up to 28 days
  Weaning period (days) between inclusion (ie first administration of loxapine/placebo) and successful extubation (no re-intubation in the following 48 hours)

SECONDARY OUTCOMES:
total duration of mechanical ventilation | up to 28 days
  -number of days of mechanical ventilation
incidence of unexpected extubations | up to 28 days
  number of patients with unexpected extubation
clinical and biological respiratory parameters | 24 hours
  description of abnormal clinical and biological respiratory parameters, number of patients concerned.
incidence of mechanical ventilation related complications | up to 48 hours after extubation
  collapses, nosocomial pneumonia, respiratory issue requiring an increase of FiO2 and/or PEP.
incidence of adverse events, related and non related to the treatment | up to 28 days
mortality rate | day 14 and week 6
  mortality rate at day 14 and week 6
factors associated to weaning failure | up to 28 days
  age, patient medical history,duration of sedation or ventilation, weaning failure

CONTACTS AND LOCATIONS:
Overall Officials: Didier Dreyfuss, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Colombes, France

REFERENCES:
- [Derived] Gaudry S, Sztrymf B, Sonneville R, Megarbane B, Van Der Meersch G, Vodovar D, Cohen Y, Ricard JD, Hajage D, Salomon L, Dreyfuss D. Loxapine to control agitation during weaning from mechanical ventilation. Crit Care. 2017 Sep 6;21(1):235. doi: 10.1186/s13054-017-1822-y. PMID 28877705